CLINICAL TRIAL: NCT02408575
Title: Hearing Aids With "Notched Amplification" for the Treatment of Chronic Tinnitus - A Controlled Randomized Pilot Study on Safety, Tolerability and Clinical Performance
Brief Title: Hearing Aids With "Notched Amplification" for the Treatment of Chronic Tinnitus
Acronym: NoA-Tin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Head of Outpatient Clinic, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Uni-Reg-NoA-Tin
Record Dates: First submitted 2015-03-18; First posted 2015-04-03 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Notched filtering (verum) (Experimental): The Hearing aid with notched amplification filters frequencies in a specific manner, depending on the individual tinnitus frequency. Through this special filtering the neuronal functional changes of the auditory cortex are supposed to be affected therapeutically.
  Intervention: Device: Conventional hearing aid type Carat 7bx with M-Receiver; Adjustment by Connexx 7.3
  Interventions: Device: Notched filtering (verum)
- No filtering (placebo) (Experimental): Conventional hearing aid type Carat 7bx with M-Receiver Adjustment by Connexx 7.3
  No notched filtering
  Intervention: Device: Conventional hearing aid type Carat 7bx with M-Receiver; Adjustment by Connexx 7.3
  Interventions: Device: No filtering (placebo)

INTERVENTIONS:
Device: Notched filtering (verum) — Conventional hearing aid type Carat 7bx with M-Receiver Adjustment by Connexx 7.3 The Hearing aid with notched amplification filters frequences in a specific manner, depending on the individual tinnitus frequency. Through this special filtering the neuronal functional changes of the auditory cortex are supposed to be affected therapeutically.
  Arms: Notched filtering (verum)
Device: No filtering (placebo) — Conventional hearing aid type Carat 7bx with M-Receiver Adjustment by Connexx 7.3
  No notched filtering
  Arms: No filtering (placebo)

SUMMARY:
Pilot study on safety, tolerability and clinical performance/randomized double-blind active-controlled pilot-study. Patients are being recruited from patients of the Tinnitus Center of Regensburg and groupwise randomized. Control groups are being treated with hearing aids without notch-filter. Patients and raters are blinded, only the coworker, who is programming the hearing aids, is informed about the group assigned.

A Hearing aid with notched amplification filters frequencies in a specific manner, depending on the individual tinnitus frequency. Through this special filtering the neuronal functional changes of the auditory cortex are supposed to be affected therapeutically.

ELIGIBILITY:
Inclusion Criteria:

* Chronic tinnitus (≥ 6 months)
* Score of ≥ 10 in TQ12 (Goebel und Hiller)
* Mild to moderate hearing loss of at least 20 dB and maximum 70 dB between 250 Hz and 8 kHz
* Tinnitus with tonal character or narrow band noise (< 1 oktave bandwidth)
* Tinnitus frequency ≤ 8 kHz in tinnitus matching
* Written informed consent of the proband
* If therapy with psychoactive substances is necessary, it has to be stable during at least 10 days and should remain constant during study (changes will be documented in the CRF)
* No regular use (8 hours daily) of hearing aids during 3 month before start of study

Exclusion Criteria:

* Objective Tinnitus
* Start of other tinnitus therapies during 3 months before start of study.
* Missing written consent
* Clinically relevant serious internal, neurologic or psychiatric diseases
* Abuse of drugs, medicaments and alcohol up to 12 weeks before start of study
* Other circumstances that object to study inclusion according to the opinion of the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mini Tinnitus Questionnaire (Mini-TQ12 of Göbel&Hiller) | Week 12
  Reduction in the sumscore means improvement of tinnitus

SECONDARY OUTCOMES:
Adverse events | Week 2
Adverse events | Week 4
Adverse events | Week 8
Adverse events | Week 12
Improvement of tinnitus measured by changes in the Tinnitus Questionnaire (TQ of Goebel&Hiller) | Week 2
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus measured by changes in the Tinnitus Questionnaire (TQ of Goebel&Hiller) | Week 4
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus measured by changes in the Tinnitus Questionnaire (TQ of Goebel&Hiller) | Week 8
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus measured by changes in the Tinnitus Questionnaire (TQ of Goebel&Hiller) | Week 12
Changes of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI of Newman et al 1996) | Week 2
  Reduction in the sumscore means improvement of tinnitus
Changes of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI of Newman et al 1996) | Week 4
  Reduction in the sumscore means improvement of tinnitus
Changes of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI of Newman et al 1996) | Week 8
  Reduction in the sumscore means improvement of tinnitus
Changes of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI of Newman et al 1996) | Week 12
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus as measured by changes in the Tinnitus Impairment Questionnaire (TBF 12) | Week 2
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus as measured by changes in the Tinnitus Impairment Questionnaire (TBF 12) | Week 4
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus as measured by changes in the Tinnitus Impairment Questionnaire (TBF 12) | Week 8
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus as measured by changes in the Tinnitus Impairment Questionnaire (TBF 12) | Week 12
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus as measured by changes in the Clinical Global Impression questionnaire (CGI) | Week 2
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus as measured by changes in the Clinical Global Impression questionnaire (CGI) | Week 4
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus as measured by changes in the Clinical Global Impression questionnaire (CGI) | Week 8
  Reduction in the sumscore means improvement of tinnitus
Improvement of tinnitus as measured by changes in the Clinical Global Impression questionnaire (CGI) | Week 12
  Reduction in the sumscore means improvement of tinnitus
Change in quality of life as measured by the WHOQoL questionnaire | Week 2
  Reduction in the sumscore means improvement of tinnitus
Change in quality of life as measured by the WHOQoL questionnaire | Week 4
  Reduction in the sumscore means improvement of tinnitus
Change in quality of life as measured by the WHOQoL questionnaire | Week 8
  Reduction in the sumscore means improvement of tinnitus
Change in quality of life as measured by the WHOQoL questionnaire | Week 12
  Reduction in the sumscore means improvement of tinnitus
Changes of tinnitus characteristics as measured by numeric rating scales (Tinnitus NRS Scales) | Week 2
  Reduction in the sumscore means improvement of tinnitus
Changes of tinnitus characteristics as measured by numeric rating scales (Tinnitus NRS Scales) | Week 4
  Reduction in the sumscore means improvement of tinnitus
Changes of tinnitus characteristics as measured by numeric rating scales (Tinnitus NRS Scales) | Week 8
  Reduction in the sumscore means improvement of tinnitus
Changes of tinnitus characteristics as measured by numeric rating scales (Tinnitus NRS Scales) | Week 12
  Reduction in the sumscore means improvement of tinnitus
Changes in psychoacoustic tinnitus characteristics | Week 2
  frequency, loudness, minimal masking level
Changes in psychoacoustic tinnitus characteristics | Week 4
  frequency, loudness, minimal masking level
Changes in psychoacoustic tinnitus characteristics | Week 8
  frequency, loudness, minimal masking level
Changes in psychoacoustic tinnitus characteristics | Week 12
  frequency, loudness, minimal masking level
Change of depressive symptoms as measured by the Major Depression Inventory (MDI) | Week 2
Change of depressive symptoms as measured by the Major Depression Inventory (MDI) | Week 4
Change of depressive symptoms as measured by the Major Depression Inventory (MDI) | Week 8
Change of depressive symptoms as measured by the Major Depression Inventory (MDI) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, M.D., Ph.D., Principal Investigator — University of Regensburg
Locations (1):
- University of Regensburg - Dept of Psychiatry and ENT Dept., Regensburg, Germany